CLINICAL TRIAL: NCT03221725
Title: The Effect of Sacrospinous Ligament Fixation After Vaginal Hysterectomy to Development of De-novo Stress Urinary Incontinence and Postoperative Vaginal Length in Treating Stage II-III Pelvic Organ Prolapse Patients
Brief Title: The Development of De-novo Stress Urinary Incontinence After Stage II-III Pelvic Organ Prolapse Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Kerem Doga Seckin, ass prof, Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016/02
Record Dates: First submitted 2017-07-14; First posted 2017-07-19 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Pelvic Organ Prolapse
Keywords: sacrospinous ligament fixation; stress urinary incontinence
MeSH Terms: conditions — Pelvic Organ Prolapse; Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- sacrospinosus fixation group (Experimental): The group which sacrospinous fixation was performed
  Interventions: Procedure: sacrospinous ligament fixation

INTERVENTIONS:
Procedure: sacrospinous ligament fixation — sacrospinous ligament fixation will be applied to prevent vaginal vault prolapse

SUMMARY:
Surgery for Stage II-III Pelvic organ prolapse

ELIGIBILITY:
Inclusion Criteria:

* Pelvic organ prolapse stage II-III
* has no incontinence before surgery

Exclusion Criteria:

* had surgery before
* Pelvic organ prolapse stage I or IV

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
development of stress urinary incontinence | in one year

SECONDARY OUTCOMES:
postoperative vaginal length | in one year

CONTACTS AND LOCATIONS:
Locations (1):
- Kerem Doga Seckin, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided